CLINICAL TRIAL: NCT04207320
Title: Hematopoietic Stem Cell Transplantation for Patients With Severe Sickle Cell Disease Using Myeloablative Conditioning and αβ+ T-cell Depleted Hematopoietic Stem Cells From Partially Matched Familial Donors
Brief Title: Haploidentical Hematopoietic Stem Cell Transplantation (HSCT) for Patients With Severe Sickle Cell Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated by PI
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-0640
Record Dates: First submitted 2019-12-11; First posted 2019-12-20 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stage I (Experimental): Stage I will include eligible subjects between the ages of 10-25 years.
  Interventions: Device: αβ+ T-cell depletion with Miltenyi CliniMACS system
- Stage II (Experimental): Stage II will include eligible subjects between the ages of 2-25 years.
  Interventions: Device: αβ+ T-cell depletion with Miltenyi CliniMACS system

INTERVENTIONS:
Device: αβ+ T-cell depletion with Miltenyi CliniMACS system — Haploidentical CD34+ megadose hematopoietic stem cell transplant in which cells are purified using the Miltenyi CliniMACS system designed for αβ+ T-cell receptor selection using immunomagnetic beads.

SUMMARY:
The purpose of this study is to develop a safe and curative stem cell transplant approach to treating sickle cell disease by assessing the safety of haploidentical hematopoietic stem cell transplantation using αβ+ T-cell depletion for children and adolescents with severe sickle cell disease (SCD).

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin SS, SC, S-β0 Thalassemia, or SO-Arab Sickle Cell Disease
* Between the ages of 2 and 25 years (Stage 1: 10-25 years; Stage II: 2-25 years)
* Lack a fully matched family donor or fully matched unrelated donor register in the National Marrow Donor Program
* Partially-matched family member with hemoglobin AA (normal) or hemoglobin AS (sickle trait) phenotype
* SCD with Severe Phenotype, defined by the following criteria: Neurologic manifestations of sickle disease including cerebral vascular accident (CVA), transient ischemic event (TIA) or abnormal MRI findings suggestive of silent infarct; Two or more episodes of acute chest syndrome (ACS) requiring admission for transfusional or respiratory support including supplemental oxygen within [two years] of enrollment in study despite hydroxyurea therapy. Patients who cannot tolerate hydroxyurea and who experience multiple episodes of ACS will also be eligible; History of severe vaso-occlusive (VOC) disease requiring hospitalization and intravenous narcotics on 3 or more occasions per year over the two years prior to enrollment despite hydroxyurea therapy. Patients who cannot tolerate hydroxyurea and who experience multiple episodes of VOC will also be eligible; Other severe phenotype as evidenced by end organ dysfunction related to sickle cell disease.

Exclusion Criteria:

* Karnofsky or Lansky score < 60%
* Acute hepatitis or evidence of moderate or severe portal fibrosis on biopsy. (Biopsy will be obtained if patient has been on chronic transfusion therapy > 6 months or has a ferritin > 1000 ng/ml) or AST or ALT >5 times the upper limit of normal
* Severe renal impairment (as evidenced by creatinine clearance of <50ml/minute glomerular filtration rate (GFR) < 50% predicted normal)
* Cardiac function that demonstrates shortening fraction less than 26% by cardiac echocardiogram or pulmonary hypertension.
* Pregnant Female.
* Lactating female.
* Pulmonary function with baseline O2 saturation <85% or Diffusing Capacity for Carbon Monoxide (DLCO) on pulmonary function testing (PFT) with a DLCO <40%.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Cunningham, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stage I | Stage II
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Stage II never opened at our site
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage I | Stage II | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 20 [16 to 22] |  | 20 [16 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety, as Measured by Incidence of Graft Failure, Grade III/IV Irreversible End Organ Toxicity, Grade III/IV aGvHD, or Death Within 100 Days Post-Hap-HSCT
Description: Graft Function: efficacy is defined as stable donor engraftment (>5% total nucleated cell DNA) and donor erythropoiesis that corrects the SCD hematologic phenotype (<50% HbS in the peripheral blood).
  Organ Toxicity: grade III/IV irreversible end organ toxicity based on NCI grading
  Graft Versus Host disease: grade III/IV aGvHD or death within 100 days post- Hap-HSCT
Time Frame: 100 days post-Hap-HSCT
Population: No subjects underwent transplant while on study. All subjects withdrawn and study closed prior to any study procedures/outcome measures performed.
Arm/Group | Stage I | Stage II
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Estimate 1-year Overall and Event-free Survival After Hap-HSCT
Description: Proportion of patients at 1 year who have not died or had graft failure
Time Frame: 1 year post transplant
Population: as for outcome 1
Arm/Group | Stage I | Stage II
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Observe the Incidence of Grades I Through IV Acute GvHD
Description: Proportion of subjects with grades I through IV acute GvHD
Time Frame: 100 days post transplant
Population: as for outcome 1
Arm/Group | Stage I | Stage II
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Observe Incidence of Severe Acute GvHD as Defined by Grades III Through IV
Description: Proportion of subjects with grades III through IV acute GvHD
Time Frame: 100 days post transplant
Population: as for outcome 1
Arm/Group | Stage I | Stage II
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Observe the Incidence of Grades I Through IV Chronic GvHD
Description: Proportion of subjects with grades I through IV chronic GvHD
Time Frame: 1 year post transplant
Population: as for outcome 1
Arm/Group | Stage I | Stage II
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Observe Incidence of Severe Chronic GvHD as Defined by Grades III and IV
Description: Proportion of subjects with grades III through IV chronic GvHD
Time Frame: 1 year post transplant
Population: as for outcome 1
Arm/Group | Stage I | Stage II
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 0 years
Description: For this Phase I study, NCI grade 1-4 AEs were to start being collected for on-study research participants from the initiation of Hydroxyurea/Azathioprine. No subject reached this point of the protocol while on study before their withdrawal. Thus, no AEs occurred for any of the three participants.
Arm/Group | Stage I | Stage II
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT04207320/Prot_SAP_000.pdf